CLINICAL TRIAL: NCT05535634
Title: Sound Ear Check (SEC) in Hearing Diagnostics in Young Children Undergoing Tympanostomy Tube Insertion
Brief Title: Sound Ear Check (SEC) in Hearing Diagnostics in Young Children
Status: Recruiting | Type: Observational
Sponsor: Vesa Lahdes (Other Government)
Responsible Party: Sponsor-Investigator, Vesa Lahdes, M.D., Turku University Hospital
Organization: Turku University Hospital (Other Government)
Other Study IDs: T9/2022
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Hearing Loss; Otitis Media With Effusion; Tympanostomy
MeSH Terms: conditions — Hearing Loss; Otitis Media with Effusion | interventions — Acoustic Impedance Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children referred for tympanostomy tube insertion: Study Sound Ear Check (SEC) hearing test among 3-10 years old otherwise healthy children referred to tympanostomy tube placement. SEC test prior surgery (with middle ear fluid) and at 1 month control visit (dry middle ear with ventilation tube). Otitis media 6 questionnaire prior surgery and at the 1 month control visit.
  Interventions: Diagnostic Test: Sound Ear Check

INTERVENTIONS:
Diagnostic Test: Sound Ear Check — Hearing test, measurement of the input impedance of the middle-ear transmission system
  Other Names: Tympanometry

SUMMARY:
Study Sound Ear Check (SEC) hearing test among 3-10 years old otherwise healthy children referred to tympanostomy tube placement. SEC test prior surgery (with middle ear fluid) and at 1 month control visit (dry middle ear with ventilation tube). Otitis media 6 questionnaire prior surgery and at the 1 month control visit.

DETAILED DESCRIPTION:
Sound Ear Check (SEC) is an automated tablet-based self-test that uses common nonspeech sounds (ecological sounds) that are accompanied by pictures that are easily recognizable even for younger children.

Before TTI operation, each participant will be tested with SEC using normal (dichotic) sounds and antiphasic sounds. Results will be compared to middle ear findings and the test will be repeated one month after the operation when the middle ears are checked to be dry (with a ventilation tube). At the time of the myringotomy during TTI operation, possible middle ear fluid will be classified as serous (transparent, clear), mucous (thick) or purulent (consisting of pus). A tympanometry will be performed within the same visit as the SEC measurement before the TTI operation. At the time of tympanometric examination, each participant will be classified as cooperative (sittings still, not crying, not resisting) or non-cooperative. Tympanometric findings will be classified after the Jerger classification. SEC and tympanometric testing is designed to be performed at the same visit as TTI operation as patients will be waiting for the operation at the ward. Medical history of the study patients will be collected from the hospital patient records and through interview and questionnaires to the subjects. Ear related quality of life questionnaire (OM-6) will be performed at the beginning of the study and the one month control visit. Questionnaires are collected using web-based REDCap -software (Research Electronic Data Capture).

ELIGIBILITY:
Inclusion Criteria:

* Finnish speaking (child and parent)

Exclusion Criteria:

* Prior sensorineural hearing loss
* developmental disorder
* Prior ear surgery (except tympanostomy insertion)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Otherwise healthy 3-10 years old children referred to tympanostomy tube insertion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
SNR | 1-2 months
  Signal to noise ratio

SECONDARY OUTCOMES:
Otitis media 6 questionnaire | 1-2 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lotta Haavisto, PhD, Principal Investigator — Hospital District of Southwest Finland
Locations (1):
- Turku University Hospital, Department of Otorhinolaryngology and head and neck surgery, Turku, Finland

IPD SHARING:
Plan to Share IPD: No